CLINICAL TRIAL: NCT04936555
Title: The Effect of Self-Acupressure Application on Functional Composite and Quality of Life in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, PhD., Assistant Prof, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 26915
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
Keywords: Self-Acupressure; Functional composite; Quality of life
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Masking Description: Self-Acupressure and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Acupressure (Experimental): Each application to the acupressure points (H17, L14, ST36, SP6) will be done in 2 minutes and right and left)
  Interventions: Other: Self-Acupressure
- No Intervention (No Intervention): Control group Routine maintenance will be applied

INTERVENTIONS:
Other: Self-Acupressure — Acupressure is a therapy method performed with an instrument or hand, fingertip, palm, elbow, knee, thumb relaxation and wrist bands on various points representing the waist organs in order to ensure the continuation and balance of the energy in our body.
  Arms: Self-Acupressure

SUMMARY:
It is important to consider the functional composite and quality of life of patients with multiple sclerosis (MS) and to plan interventions for these problems.

DETAILED DESCRIPTION:
The application of Self-Acupressure helps in improving the functional composite and quality of life in Multiple Sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* To be able to communicate adequately
* Not having psychiatric problems
* Volunteering to participate in research

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Multiple Sclerosis Functional Composite (MSFC) | 1. week
  The conventional MSFC battery (MSFC3), comprising the 25 foot timed walk test (TWT), 9-hole peg test (9HPT) and paced auditory serial addition test (PASAT) was performed according to standardised procedures, calculated according to the standard manual, and normalised to this cohort.
Multiple Sclerosis Functional Composite (MSFC) | 4. week
  The conventional MSFC battery (MSFC3), comprising the 25 foot timed walk test (TWT), 9-hole peg test (9HPT) and paced auditory serial addition test (PASAT) was performed according to standardised procedures, calculated according to the standard manual, and normalised to this cohort.
Multiple Sclerosis Quality of Life Scale-54 | 1.week
  This scale was developed by Vickrey et al17 to evaluate the quality of life of patients with The scale was created by adding 18 MS-related items to SF-36 (short form). Physical and mental health composite scores are calculated, and higher scores indicate better quality of life. The Turkish version was developed by Tulek et al.
Multiple Sclerosis Quality of Life Scale-54 | 4.week
  This scale was developed by Vickrey et al17 to evaluate the quality of life of patients with The scale was created by adding 18 MS-related items to SF-36 (short form). Physical and mental health composite scores are calculated, and higher scores indicate better quality of life. The Turkish version was developed by Tulek et al.

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz ÖZER, PhD, Study Chair — Istanbul Sabahattin Zaim University
Locations (1):
- Istanbul Sabahattin Zain Universitiy, Istanbul, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bastani F, Sobhani M, Emamzadeh Ghasemi HS. Effect of acupressure on fatigue in women with multiple sclerosis. Glob J Health Sci. 2015 Jan 26;7(4):375-81. doi: 10.5539/gjhs.v7n4p375. PMID 25946938